CLINICAL TRIAL: NCT01415544
Title: An Evaluation and Comparison of Noninvasive Blood Glucose Concentrations Relative to Finger Capillary Blood Glucose References
Brief Title: Comparison of Noninvasive Blood Glucose Concentrations Relative to Finger Capillary Blood Glucose References
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: InLight Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-0020
Record Dates: First submitted 2011-08-09; First posted 2011-08-12 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Gestational Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — capillary glucose measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Type 2 Diabetes: Those previously diagnosed with type 2 diabetes
- Type 1 Diabetes: Those previously diagnosed with type 1 diabetes
- Gestational Diabetes: Those that are currently diagnosed with gestational diabetes
- Healthy Human Volunteers: Those that have not been diagnosed with any type of diabetes

SUMMARY:
The purpose of the study is to prospectively evaluate a noninvasive, near-infrared based method for measuring glucose concentration relative to invasive blood reference measurements. The initial phase of the study will be focused on procurement of the data needed to develop a robust, accurate calibration. The second phase will be focused on performance evaluation of the system.

DETAILED DESCRIPTION:
Currently, individuals with diabetes must use an invasive finger stick methodology for the determination of their blood glucose levels. Although current technology glucose meters use a smaller amount of blood than older generation meters, the pain and inconvenience associated with this invasive measurement is the number one reason cited for inadequate or infrequent blood glucose monitoring. In fact up to 67% of patients with diabetes fail to routinely monitor their blood glucose levels. A survey of 1895 patients showed that finger soreness was the most common reason given for self-reported noncompliance with testing recommendations, followed by pain, inconvenience, fear of needles, and "other" (including cost), (Diabetes Care August 2001 vol. 24 no. 8 1502-1503). The ability to make a painless blood glucose measurement using only light would address the pain and inconvenience issues associated with current technology glucose meters.

The initial application of the technology is associated with the monitoring of Gestational Diabetes. The International Association of Diabetes and Pregnancy Study Groups (IADPSG) recently released recommendations for diagnosing gestational diabetes, as well as clarifying the benefits of treatment (Diabetes Care, 2010;33:676-682). The IADPSG cited research that found significant graded relationships between increasing maternal glucose levels and the frequency of four primary and five secondary outcomes. For example, with a 1-standard deviation increase in maternal fasting, 1-hour, and 2-hour plasma glucose levels, there was a corresponding 38%, 46%, and 38% increased risk, respectively, in the primary outcome of birth weight >90th percentile, and a 5%, 18%, and 16% increased risk, respectively, of the secondary outcome of premature delivery before 37 weeks gestation (N Engl J Med 2008;358:1991-2002).

ELIGIBILITY:
Inclusion Criteria:

* Female at least 20 years of age but not older than 50 years of age
* Female with Type I or Gestational diabetes based on ADA criteria
* Female with Type II diabetes and A1c of greater than 7.0 as measured on a Bayer A1C Now meter
* May include female healthy volunteers.

Exclusion Criteria:

* Subject requires hemo-dialysis
* Severe heart disease as evidenced by peripheral edema
* Liver disease as evidenced by jaundice
* Active alcohol or drug abuse
* Body Mass Index (BMI) > 35 kg/m2
* Hand size too large to fit in the optical measurement instrumentation
* Middle finger width of less than 5 mm
* Skin damage at optical sampling site on hand
* Currently taking prednisone or other systemic steroids
* Tattoo at the optical sampling site

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Human Subject population consists of female subjects between the ages of 20 and 50. Subjects must have been diagnosed with either Type I, Type II, or Gestational diabetes and may utilize healthy individuals for the validation phase. Up to 100 subjects may be recruited to participate in this study. Subjects will be recruited from the community and will be selected to ensure a representative sample of the projected intended use population. Efforts will also be made to ensure a broad and even distribution of ages (between 20 and 50 years old) and ethnicities.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Calibrate near-infrared spectroscopy-based glucose meter | 1 year
  The collection of capillary blood glucose and noninvasive data will allow the calibration of the noninvasive systems and subsequently evaluate performance via a validation study. The paired NIR spectrum and blood reference data acquired during calibration will be processed using multivariate regression techniques to create a calibration model. Results will be compared using a Clark error grid.

SECONDARY OUTCOMES:
Compare Noninvasive to invasive techniques | 1 year
  Comparison of noninvasive glucose measurement performance versus standard invasive reference. Invasive measurements are made by obtaining capillary blood glucose measurements and then measuring blood on a Yellow Springs Instrument (YSI). Due to the fact that instrumentation drift and subject physiological changes can adversely influence measurement performance, the study is specifically designed to examine performance over an appropriate period of time with a reasonable distribution of subject variance. Results will be compared using a Clark error grid.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Forman, MD, Principal Investigator — Lovelace Scientific Resources
Locations (1):
- Lovelace Scientific Resources, Albuquerque, New Mexico, United States